CLINICAL TRIAL: NCT04570306
Title: Whole Blood Transcriptional and Mass Cytometry Immune Profiling in Systemic Lupus Erythematosus (SLE) Patients to Discern the Salutary Effects of Belimumab on Halting Disease Progression and Flares Without Compromising Host Fitness
Brief Title: Transcriptional and Immune Parameters of Response to Belimumab
Status: Completed | Type: Observational
Sponsor: Biomedical Research Foundation, Academy of Athens (Other)
Collaborators: Attikon Hospital (Other); University Hospital of Heraklion (Unknown); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, DIMITRIOS BOUMPAS, Professor and Chairman Department of Medicine, Medical School, National and Kapodestrian University of Athens, Biomedical Research Foundation, Academy of Athens
Other Study IDs: DB11
Record Dates: First submitted 2020-06-19; First posted 2020-09-30 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Systemic Lupus Erythematosus
Keywords: transcriptome; trained immunity; host-pathogen defense
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood RNA tubes, ethylenediaminetetraacetic acid (EDTA) tubes for genomic DNA extraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Belimumab-treated SLE patients: SLE patients with active disease who will be started on add-on treatment with belimumab on top of standard of care.
  Interventions: Drug: Belimumab

INTERVENTIONS:
Drug: Belimumab — The study will involve 80 adult patients diagnosed with SLE who will be started on belimumab (standard approved dose of i.v. 10 mg/kg or subcutaneous 200 mg/week) due to active disease. The intention to start belimumab will be made by the treating Rheumatologist(s), in accordance to the current standard of care, and on the basis of shared physician-patient decision making.

SUMMARY:
The investigators propose to perform RNA-sequencing of the whole blood initially, in a cohort of 80 SLE patients who will receive belimumab as part of standard clinical practice, in order to assess intra-patient longitudinal (baseline, 1, 3 and 6 months) transcriptome changes and examine whether treatment can ameliorate the activity/flare, severity and major organ disease gene signatures. The investigators will also obtain preliminary information on molecular signatures predicting clinical responses and the impact of belimumab on gene signatures of host defense against viral and bacterial (including mycobacterial) pathogens. Using modules of cell type-specific genes and co-expression gene networks, The investigators will deconvolute our data to define pertinent molecular alterations in specific immune cell types. Results will be validated and functionally characterized by single-cell mass cytometry (performed at the aforementioned time points), which enables investigation of the cell identity (including subsets of B-cells and myeloid cells of particular relevance to the disease) and activation status at protein level (e.g. phosphorylation) through next-generation, high-dimensional flow cytometry. Through a focused analysis followed by targeted gene expression and function studies in purified monocytes, the investigators will determine whether belimumab can restore "SLE-primed" monocytes thus, alleviating their inflammatory and pro-atherogenic phenotype and enhancing their bactericidal activity. Collectively, these studies will provide novel mechanistic insights on the beneficial efficacy/toxicity ratio of belimumab therapy in SLE.

DETAILED DESCRIPTION:
B-cell activating factor (BAFF) excess causes lupus disease by exerting costimulatory effects on the B-cell compartment but also on a variety of non-B-cell subsets such as T-helper cells and monocytes/dendritic cells. The 2019 updated European League Against Rheumatism (EULAR) recommendations for SLE recommend usage of belimumab (anti-BAFF mAb) in persistently active or flaring disease based upon evidence for efficacy, reduction of flares and organ damage accrual without increasing the risk of infections. Still, belimumab is usually reserved for established, refractory cases. It is conceivable that earlier usage may halt the progression of the disease, especially prevent flares and dysfunction in major organs. The investigators have completed a combined genetic and transcriptomic analysis in the peripheral blood of SLE patients and have characterized distinct gene signatures for disease activity/flare and severity. Using machine learning techniques, the investigators can predict SLE patients likely to develop major organ involvement. In vitro and gene profiling studies in purified lupus monocytes indicate that these cells exist - under the effect of type I interferon - in a "high alert" autoreactive and metabolic state (reminiscent of 'trained immunity'), which may contribute to risk of flares, tissue injury but also major comorbidities seen in SLE, particularly accelerated atherosclerosis and infections. Based upon the clinical experience accumulated thus far, it is likely that belimumab may neutralize these molecular signatures for flares and disease progression without interfering with host defense immune pathways.

The investigators propose to perform RNA-sequencing of the whole blood initially, in a cohort of 80 SLE patients who will receive belimumab as part of standard clinical practice, in order to assess intra-patient longitudinal (baseline, 1, 3 and 6 months) transcriptome changes and examine whether treatment can ameliorate the identified activity/flare, severity and major organ disease signatures. The investigators will also obtain preliminary information on molecular signatures predicting clinical responses and the impact of belimumab on gene signatures of host defense against viral and bacterial (including mycobacterial) pathogens. Using modules of cell type-specific genes and co-expression gene networks, the investigators will deconvolute our data to define pertinent molecular alterations in specific immune cell types. Results will be validated and functionally characterized by single-cell mass cytometry (performed at the aforementioned time points), which enables investigation of the cell identity (including subsets of B-cells and myeloid cells of particular relevance to the disease) and activation status at protein level (e.g. phosphorylation) through next-generation, high-dimensional flow cytometry. Through a focused analysis of the deconvoluted RNA-seq and mass cytometry data followed by targeted gene expression and function studies in purified monocytes, the investigators will determine whether belimumab can restore "SLE-primed" monocytes thus, alleviating their inflammatory and pro-atherogenic phenotype and enhancing their bactericidal activity. Collectively, these studies will provide novel mechanistic insights on the beneficial efficacy/toxicity ratio of belimumab therapy in SLE, while supporting the early use of the drug.

ELIGIBILITY:
Inclusion Criteria: SLE patients:

* who meet the Systemic Lupus International Collaborating Clinics (SLICC) 2012 and/or European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) 2019 classification criteria;
* have active disease defined as the combination of clinical (i.e., excluding serology) SLEDAI-2000 ≥6 and/or physician global assessment (PhGA) ≥1.5. Both flaring (acute exacerbation) and persistent disease activity will be considered;
* are started belimumab (standard approved dose of i.v. 10 mg/kg or subcutaneous 200 mg/week) due to active disease. The intention to start belimumab will be made by the treating Rheumatologist(s), in accordance to the current standard of care, and on the basis of shared physician-patient decision making.

Exclusion Criteria:

* age <18 years
* co-existing rheumatic or other autoimmune disease
* pregnancy
* active infection
* history of malignant disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will involve 80 adult patients diagnosed with SLE (according to the SLICC 2012 and/or EULAR/ACR 2019 classification criteria) who will be started on belimumab (standard approved dose of i.v. 10 mg/kg or subcutaneous 200 mg/week) due to active disease. The intention to start belimumab will be made by the treating Rheumatologist(s), in accordance to the current standard of care, and on the basis of shared physician-patient decision making. Active SLE is defined as the combination of clinical (i.e., excluding serology) SLEDAI-2K ≥6 and/or physician global assessment (PhGA) ≥1.5. Both flaring (acute exacerbation) and persistent disease activity will be considered.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2023-12-16 (Actual); Study Completion 2023-12-16 (Actual)

PRIMARY OUTCOMES:
Changes in blood transcriptome in relation to clinical response induced by belimumab | 1, 3 and 6 months
  To evaluate changes in SLE blood transcriptome that are induced by treatment with belimumab with emphasis on the reversibility of previously-defined gene signatures for disease activity/flare, severity/progression and major organ involvement. Results will be correlated with validated patient outcomes such as clinical response (defined according to SLE Responder Index-4).

SECONDARY OUTCOMES:
Changes in blood transcriptome in relation to low disease activity induced by belimumab | 3 and 6 months
  To evaluate changes in SLE blood transcriptome that are induced by treatment with belimumab with emphasis on the reversibility of previously-defined gene signatures for disease activity/flare, severity/progression and major organ involvement. Results will be correlated with low disease activity in SLE (according to the Low Disease Activity State definition)
Changes in blood transcriptome in relation to remission induced by belimumab | 6 months
  To evaluate changes in SLE blood transcriptome that are induced by treatment with belimumab with emphasis on the reversibility of previously-defined gene signatures for disease activity/flare, severity/progression and major organ involvement. Results will be correlated with remission in SLE (according to the Definition of Remission [DORIS] in SLE)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios T Boumpas, MD, Study Chair — Biomedical Research Foundation, Academy of Athens
Locations (1):
- BRFAA, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Steri M, Orru V, Idda ML, Pitzalis M, Pala M, Zara I, Sidore C, Faa V, Floris M, Deiana M, Asunis I, Porcu E, Mulas A, Piras MG, Lobina M, Lai S, Marongiu M, Serra V, Marongiu M, Sole G, Busonero F, Maschio A, Cusano R, Cuccuru G, Deidda F, Poddie F, Farina G, Dei M, Virdis F, Olla S, Satta MA, Pani M, Delitala A, Cocco E, Frau J, Coghe G, Lorefice L, Fenu G, Ferrigno P, Ban M, Barizzone N, Leone M, Guerini FR, Piga M, Firinu D, Kockum I, Lima Bomfim I, Olsson T, Alfredsson L, Suarez A, Carreira PE, Castillo-Palma MJ, Marcus JH, Congia M, Angius A, Melis M, Gonzalez A, Alarcon Riquelme ME, da Silva BM, Marchini M, Danieli MG, Del Giacco S, Mathieu A, Pani A, Montgomery SB, Rosati G, Hillert J, Sawcer S, D'Alfonso S, Todd JA, Novembre J, Abecasis GR, Whalen MB, Marrosu MG, Meloni A, Sanna S, Gorospe M, Schlessinger D, Fiorillo E, Zoledziewska M, Cucca F. Overexpression of the Cytokine BAFF and Autoimmunity Risk. N Engl J Med. 2017 Apr 27;376(17):1615-1626. doi: 10.1056/NEJMoa1610528. PMID 28445677
- [Background] Kang S, Fedoriw Y, Brenneman EK, Truong YK, Kikly K, Vilen BJ. BAFF Induces Tertiary Lymphoid Structures and Positions T Cells within the Glomeruli during Lupus Nephritis. J Immunol. 2017 Apr 1;198(7):2602-2611. doi: 10.4049/jimmunol.1600281. Epub 2017 Feb 24. PMID 28235864
- [Background] Urowitz MB, Ohsfeldt RL, Wielage RC, Kelton KA, Asukai Y, Ramachandran S. Organ damage in patients treated with belimumab versus standard of care: a propensity score-matched comparative analysis. Ann Rheum Dis. 2019 Mar;78(3):372-379. doi: 10.1136/annrheumdis-2018-214043. Epub 2019 Jan 4. PMID 30610066
- [Background] Panousis NI, Bertsias GK, Ongen H, Gergianaki I, Tektonidou MG, Trachana M, Romano-Palumbo L, Bielser D, Howald C, Pamfil C, Fanouriakis A, Kosmara D, Repa A, Sidiropoulos P, Dermitzakis ET, Boumpas DT. Combined genetic and transcriptome analysis of patients with SLE: distinct, targetable signatures for susceptibility and severity. Ann Rheum Dis. 2019 Aug;78(8):1079-1089. doi: 10.1136/annrheumdis-2018-214379. Epub 2019 Jun 5. PMID 31167757
- [Background] Novakovic B, Habibi E, Wang SY, Arts RJW, Davar R, Megchelenbrink W, Kim B, Kuznetsova T, Kox M, Zwaag J, Matarese F, van Heeringen SJ, Janssen-Megens EM, Sharifi N, Wang C, Keramati F, Schoonenberg V, Flicek P, Clarke L, Pickkers P, Heath S, Gut I, Netea MG, Martens JHA, Logie C, Stunnenberg HG. beta-Glucan Reverses the Epigenetic State of LPS-Induced Immunological Tolerance. Cell. 2016 Nov 17;167(5):1354-1368.e14. doi: 10.1016/j.cell.2016.09.034. PMID 27863248
- [Background] van Vollenhoven RF, Petri MA, Cervera R, Roth DA, Ji BN, Kleoudis CS, Zhong ZJ, Freimuth W. Belimumab in the treatment of systemic lupus erythematosus: high disease activity predictors of response. Ann Rheum Dis. 2012 Aug;71(8):1343-9. doi: 10.1136/annrheumdis-2011-200937. Epub 2012 Feb 15. PMID 22337213
- [Background] Goh C, Knight JC. Enhanced understanding of the host-pathogen interaction in sepsis: new opportunities for omic approaches. Lancet Respir Med. 2017 Mar;5(3):212-223. doi: 10.1016/S2213-2600(17)30045-0. PMID 28266329
- [Background] Monaco G, Lee B, Xu W, Mustafah S, Hwang YY, Carre C, Burdin N, Visan L, Ceccarelli M, Poidinger M, Zippelius A, Pedro de Magalhaes J, Larbi A. RNA-Seq Signatures Normalized by mRNA Abundance Allow Absolute Deconvolution of Human Immune Cell Types. Cell Rep. 2019 Feb 5;26(6):1627-1640.e7. doi: 10.1016/j.celrep.2019.01.041. PMID 30726743